CLINICAL TRIAL: NCT04008875
Title: Improvement of Weaning From Mechanical Ventilation by Continuous Ultrasound Monitoring of Diaphragm Excursion: the WEAN-US Study
Brief Title: Improvement of Weaning From Mechanical Ventilation by Continuous Ultrasound Monitoring of Diaphragm Excursion
Acronym: WEAN-US
Status: Completed | Type: Observational
Sponsor: Respinor AS (Industry)
Collaborators: European Commission (Other)
Responsible Party: Sponsor
Other Study IDs: DM-CS-003
Record Dates: First submitted 2019-04-12; First posted 2019-07-05 (Actual); Last update posted 2021-06-14 (Actual); Status verified 2021-06

CONDITIONS: Respiration, Artificial
Keywords: diaphragm ultrasound; mechanical ventilation; diaphragm function
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Successful weaning/extubation: Successful weaning will be defined as a patient who completes a planned 30-minute spontaneous breathing trial.
  Successful extubation will be defined as a patient who completes a planned 30-minute spontaneous breathing trial and is not reintubated in the first 48 hours after extubation.
- Failed weaning/extubation: Failed weaning will be defined as a patient who did not complete a planned 30-minute spontaneous breathing trial.
  Failed extubation will be defined as a patient who did not complete a planned 30-minute spontaneous breathing trial, in the first 48 hours after extubation are reintubated, have unplanned non-invasive ventilation (NIV) or who have a tracheostomy.

SUMMARY:
Justification: The diaphragm is the main inspiratory muscle. Its dysfunction therefore compromises ventilation, which is necessary for gas exchange. Diaphragmatic dysfunction is frequently observed in resuscitation patients. Diaphragm ultrasound is currently a simple and validated technique for measuring the function of the diaphragm in intensive care. However, the discontinuity of the measurements is one of the major limitations of the current, standard ultrasonic evaluation of diaphragm function. Respinor AS (Oslo, Norway) has developed an ultrasound device (known as RESPINOR DXT) for continuous quantification of diaphragmatic excursion and velocity.

Aims of the study: To evaluate the feasibility of the continuous monitoring of the diaphragmatic excursion using RESPINOR DXT in patients undergoing MV in the intensive care unit, to ensure its reliability and to establish a link between the diaphragmatic excursion and the weaning outcome of MV.

Method: In addition to continuous diaphragm monitoring by RESPINOR DXT, a daily measurement of the diaphragm excursion will be performed using a conventional ultrasound system for comparison. A daily measurement of the oesophageal pressure (Pes) and the gastric pressure (Pga) will be performed, thus allowing the calculation of the transdiaphragmatic pressure (Pdi).

Analysis: The feasibility of the measurement will be evaluated through user utility questions as well as the time spent with a signal meeting specific quality criteria. Its reliability will be studied by the concordance between the measurements of the excursion measured by RESPINOR DXT and by standard ultrasound (Bland-Altman, Passing-Bablock). It will be further evaluated by the correlation between the variations of the excursion measured by RESPINOR DXT and the Pdi variations. Receiver operating characteristic (ROC) curves will be performed to identify the optimal diaphragmatic excursion threshold for predicting weaning success and prognosis.

Hypothesis: It is anticipated that the present study will show that the continuous monitoring of diaphragm excursion by RESPINOR DXT is reliable. Further, it is anticipated that there will be a statistical link between the diaphragmatic excursion and velocity of the movement measured by RESPINOR DXT before, during and after the spontaneous breathing trial.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old
* Consent to participate in the study
* Affiliation to a social security scheme or entitled to it
* Invasive mechanical ventilation for ≥ 24 hours
* Richmond Agitation Sedation Scale (RASS) ≥ - 3 (Moderate sedation)
* Able to tolerate spontaneous ventilation with inspiratory support ≤ 28 cmH2O
* Absence of high-dose vasopressors defined by noradrenaline dosage < 0.3 μg / kg / min

Exclusion Criteria:

* Central or spinal neurological lesion involving central ventilatory control or its transmission
* Contraindication to the insertion of the oesophageal catheter, ie any contraindication to insertion or change of gastric tube, esophageal surgery of less than 14 days, oesophageal varices rupture of less than 4 days
* Known neuromuscular disease, curare less than 24 hours (excluding succinylcholine for rapid sequence intubation), known hemidiaphragm paralysis or suspicion of hemidiaphragm paralysis (defined by elevation) dome> 2.5 cm compared to contralateral dome
* Patient in therapeutic limitation
* Pregnant woman, minor patient or protected adult

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients on mechanical ventilation in the intensive care unit for greater than 24 hours
Sampling Method: Non-Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2019-04-11 (Actual); Primary Completion 2020-07-08 (Actual); Study Completion 2020-10-14 (Actual)

PRIMARY OUTCOMES:
User-completed 5-point utility questions | Day 1 of enrolment
  Five-point scale to assess ease of application of the device. Scale used has options of very difficult, difficult, neutral, easy, very easy, with very easy being the better outcome and very difficult the worst.
Incidence of pressure sores. | Up to 14 days (the period of enrolment of the patient)
  The investigators will measure the incidence of pressure sores at the site of the investigative device sensors in patients throughout the period of enrolment.

SECONDARY OUTCOMES:
Concordance between diaphragm excursion measurements. | Up to 14 days (the period of enrolment of the patient)
  Comparison with a "gold standard". Concordance between diaphragm excursion measurements measured by the RESPINOR DXT monitor and standard ultrasound will be assessed using Bland-Altman analysis.
Changes in diaphragm excursion during the SBT. | From 30 minutes before the SBT up to 30 minutes post-SBT
  Receiver operating characteristic (ROC) curves will be performed to identify the optimal diaphragmatic excursion threshold for predicting weaning success.
Correlation between the diaphragm velocity and transdiaphragmatic pressure measurements. | From 30 minutes before the SBT up to 30 minutes post-SBT
  Correlations between diaphragm velocity measured by the RESPINOR DXT and the Pdi variations measured by the orogastric catheter will be made.

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Demoule, MD, Principal Investigator — Hôpital Universitaire Pitié Salpêtrière
Locations (3):
- France (3):
  - CHU Angers, Angers
  - CH Saint Joseph Saint Luc, Lyon
  - Hôpital Universitaire Pitié Salpêtrière, Paris

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Jiang JR, Tsai TH, Jerng JS, Yu CJ, Wu HD, Yang PC. Ultrasonographic evaluation of liver/spleen movements and extubation outcome. Chest. 2004 Jul;126(1):179-85. doi: 10.1378/chest.126.1.179. PMID 15249460
- [Background] Spadaro S, Grasso S, Mauri T, Dalla Corte F, Alvisi V, Ragazzi R, Cricca V, Biondi G, Di Mussi R, Marangoni E, Volta CA. Can diaphragmatic ultrasonography performed during the T-tube trial predict weaning failure? The role of diaphragmatic rapid shallow breathing index. Crit Care. 2016 Sep 28;20(1):305. doi: 10.1186/s13054-016-1479-y. PMID 27677861
- [Background] Jaber S, Petrof BJ, Jung B, Chanques G, Berthet JP, Rabuel C, Bouyabrine H, Courouble P, Koechlin-Ramonatxo C, Sebbane M, Similowski T, Scheuermann V, Mebazaa A, Capdevila X, Mornet D, Mercier J, Lacampagne A, Philips A, Matecki S. Rapidly progressive diaphragmatic weakness and injury during mechanical ventilation in humans. Am J Respir Crit Care Med. 2011 Feb 1;183(3):364-71. doi: 10.1164/rccm.201004-0670OC. Epub 2010 Sep 2. PMID 20813887
- [Background] Levine S, Nguyen T, Taylor N, Friscia ME, Budak MT, Rothenberg P, Zhu J, Sachdeva R, Sonnad S, Kaiser LR, Rubinstein NA, Powers SK, Shrager JB. Rapid disuse atrophy of diaphragm fibers in mechanically ventilated humans. N Engl J Med. 2008 Mar 27;358(13):1327-35. doi: 10.1056/NEJMoa070447. PMID 18367735
- [Background] Kim WY, Suh HJ, Hong SB, Koh Y, Lim CM. Diaphragm dysfunction assessed by ultrasonography: influence on weaning from mechanical ventilation. Crit Care Med. 2011 Dec;39(12):2627-30. doi: 10.1097/CCM.0b013e3182266408. PMID 21705883
- [Background] Llamas-Alvarez AM, Tenza-Lozano EM, Latour-Perez J. Diaphragm and Lung Ultrasound to Predict Weaning Outcome: Systematic Review and Meta-Analysis. Chest. 2017 Dec;152(6):1140-1150. doi: 10.1016/j.chest.2017.08.028. Epub 2017 Aug 31. PMID 28864053
- [Background] Zambon M, Greco M, Bocchino S, Cabrini L, Beccaria PF, Zangrillo A. Assessment of diaphragmatic dysfunction in the critically ill patient with ultrasound: a systematic review. Intensive Care Med. 2017 Jan;43(1):29-38. doi: 10.1007/s00134-016-4524-z. Epub 2016 Sep 12. PMID 27620292
- [Background] Farghaly S, Hasan AA. Diaphragm ultrasound as a new method to predict extubation outcome in mechanically ventilated patients. Aust Crit Care. 2017 Jan;30(1):37-43. doi: 10.1016/j.aucc.2016.03.004. Epub 2016 Apr 22. PMID 27112953
- [Derived] Demoule A, Fosse Q, Mercat A, Bergum D, Virolle S, Bureau C, Mellemseter M, Guichou R, Similowski T, Dres M, Mortaza S. Operator independent continuous ultrasound monitoring of diaphragm excursion predicts successful weaning from mechanical ventilation: a prospective observational study. Crit Care. 2024 Jul 16;28(1):245. doi: 10.1186/s13054-024-05003-0. PMID 39014512